CLINICAL TRIAL: NCT02499861
Title: A Phase I/IIa Study of Decitabine in Combination With Genistein in Pediatric Patients With Relapsed or Refractory Solid Tumors and Leukemia
Brief Title: Phase I/II a Study of Decitabine in Combination With Genistein in Pediatric Relapsed or Refractory Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Henrique Bittencourt, MD, PhD, Pediatric Hematologist-Oncologist, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEC-GEN001
Record Dates: First submitted 2015-02-10; First posted 2015-07-16 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Decitabine; Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine and Genistein (Experimental): continuous 24 hours Intravenous decitabine followed by oral genistein for 20 days.
  Interventions: Drug: Decitabine and Genistein

INTERVENTIONS:
Drug: Decitabine and Genistein — intravenous Decitabine with oral genistein

SUMMARY:
This Phase I/IIa study will test the combination of the epigenetic drug decitabine with the isoflavone genistein in children with leukemias and solid tumors. For the phase I study, the maximum tolerated dose will be evaluated in pediatric patients with relapsed or refractory leukemia and solid tumors. For the phase II study, only patients with relapsed or refractory leukemias will be included. To further evaluate the treatment efficacy and gain further insight into action of these drugs, the DNA methylation levels before and after treatment for all participants, pharmacokinetics parameters such as through level for decitabine and through and peak level for genistein will be measured. Pharmacogenomics testing for decitabine will be performed prior to cycle 1 of treatment.

Decitabine will be administered over a 24 hours infusion on day 1 of cycle (28 days) and genistein will be taken orally twice daily from day 2 to 21, followed by a 7 days rest period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years of age and < 21 years of age at time of study enrollment
* Able to swallow genistein or take it with a puree.
* Patients must have a diagnosis of recurrent or refractory solid tumors, including Central Nervous System tumors, lymphoma or leukemia for which standard curative measures do not exist or are no longer effective
* For solid tumors, patients must have either measurable or evaluable disease. For leukemia, patients must have > 5% blasts in the bone marrow.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy.
* Performance level: Karnofsky ≥50% for patients ≥ 16 years of age or Lansky ≥ 50% for patients < 16 years of age
* Life expectancy at least one month
* Patients must have adequate bone-marrow function
* Patients must have normal organ as defined below: (total bilirubin ≤ 24microM/L), Amylase/pancreatic amylase≤1.5 × institutional upper limit of normal, Aspartate Aminotransferase (AST) /Alanine Aminotransferase (ALT) ≤2.5 × institutional upper limit of normal, creatinine clearance ≥60 mL/min/1.73 m2.

OR creatinine according to age/gender

* Nervous system disorders (CTCAE v4) resulting from prior therapy must be ≤ Grade 2
* Participants of child-bearing potential and men must agree to use adequate contraception for the duration of study treatment, and 4 months after completion of decitabine and genistein administration.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent

Exclusion Criteria:

* Prior decitabine or genistein therapy.
* Patients who are receiving any other investigational agents.
* Nasogastric or gastrostomy (or equivalent) administration of genistein is not allowed.
* Patients with known exclusive non-measurable leptomeningeal disease at enrolment should be excluded from this clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine and genistein.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (receiving antibiotics), symptomatic heart or lung disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast-feeding women are excluded from this study. All girls of child bearing potential must have a negative pregnant test prior to enrolment.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of the combination of intravenous decitabine with oral genistein for children with refractory or recurrent solid malignancies and leukemia | 12-18 mnths
Number of participants with adverse events as a measurement of safety and tolerability of the combination of intravenous decitabine with oral genistein in children. | 12-18 months
Clinical benefit of the combination of intravenous decitabine with oral genistein in phase IIa of the study measure by either volumetric MRI for solid tumor or by bone marrow aspiration or biopsy for leukemia) at the end of cycle 2, 4, 6, 9 and 12. | 42 months

SECONDARY OUTCOMES:
Plasma concentration of decitabine and genistein during cycle 1 and 2 (just in Phase I). | 12-18 months
DNA methylation levels in selected gene promoters before and after treatment. | 42 months
Quality of life assess through Peds Quality of Life Cancer module, Peds Quality of Life Fatigue module, Reported Health status 15-items, Pain Visual Analogue Scale, Distress Rating Scale, Expectations and McGill Quality of Life Questionnaire | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Bittencourt, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada